CLINICAL TRIAL: NCT06341387
Title: Volatolomic and Proteomic Profile; Breath, Urine and Serum as Non-invasive Tools for Early Diagnosis of Lung Cancer
Brief Title: Volatolomic and Proteomic Profile for Early Diagnosis of Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Collaborators: University of Rome Tor Vergata (Other)
Responsible Party: Sponsor
Other Study IDs: R178522-ieo1906
Record Dates: First submitted 2024-03-18; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2023-10

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer Stage I; Non-small Cell Lung Cancer Stage II; Lung Cancer Diagnosis
Keywords: Lung cancer; early diagnosis; Biomarkers; Proteomic; Volatomic
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Disease | interventions — Urination; Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples Without DNA — serum samples urine samples exhaled breath samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lung cancer patients: Age 50-80 years Diagnosis of early stage of lung cancer No previous chemo or radiotherapy for lung cancer No previous malignancies within last 5 years No abuse of alcohol (no more than 1 litre of wine for day). No patients with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study Signed Informed Consent Completed questionnaire
  Interventions: Other: Breath, urine and blood analysis
- High Risk-Healthy Subjects: Age 50-80 years high risk individuals (heavy smokers, subjects with pulmonary disease non-cancer related or with a familiar history of lung cancer disease) Recent (within 6 months) negative Chest X-ray or CT scan No previous malignancies within last 5 years No patients with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study Signed Informed Consent Completed questionnaire
  Interventions: Other: Breath, urine and blood analysis

INTERVENTIONS:
Other: Breath, urine and blood analysis — breath sampling: all subjects exhale into two sterile Tedlar bags, connected to a mouthpiece, in a condition similar to traditional spirometry.
  Urine will be collected usual urine container.
  The blood sample (~ 5 ml) will be taken with a serum separator tube.

SUMMARY:
The goal of this prospective, case-control study is to discover the specific "omics" biomarkers of early stage of lung cancer using the non-invasive samples (breath, urine and serum) in a total of 200 subjects (100 healthy controls and 100 lung cancer patient). The main questions it aims to answer are:

* Which are the "omics" biomarkers that characterize the early stage of lung cancer?
* How to Translate Laboratory Data into Clinical Data?

For each participant we will collected the breath, urine and blood samples. In lung cancer patients group the samples will be sample before lung cancer resection. The samples of Breath, urine and serum will be analysed using different type of analysis: eNose and the Gas Chromatography combined with Ion Mass Spectrometry (GC/IMS). Moreover, Serum will be analyzed by mass-spectrometry-based proteomics. The purpose of these analyses will be to find biomarkers capable of distinguishing the early-stage of lung cancer from the healthy group. Followup will be performed to evaluate the possible change of the volatolomic and proteomic profile.

DETAILED DESCRIPTION:
All partecipants will sign the Informed Consent before the sampling procedures. In addition, they will complete the clinical questionnaire containing medical history, smoking history and psychological evaluation.We will conduct the trial according to the ICH Good Clinical Practice (GCP) guidelines. Keeping accurate and consistent records is essential to a cooperative study.The IEO Data Management Office will responsible of the study database and data management.

ELIGIBILITY:
Inclusion Criteria:

1. Lung cancer group

   * Diagnosis of early stage - lung cancer
   * Signed Informed Consent
   * Completed questionnaire
2. Healthy subjects

   * high risk individuals (heavy smokers, subjects with pulmonary disease non-cancer related or with a familiar history of lung cancer disease)
   * Recent (within 6 months) negative Chest X-ray or CT scan

Exclusion Criteria:

Both groups

* No previous chemo or radiotherapy for lung cancer
* No previous malignancies within last 5 years
* No abuse of alcohol (no more than 1 litre of wine for day).
* No patients with psychiatric, addictive, or any disorder, which compromises ability to give informed consent for participation in this study

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Our experimental design consists to submit two groups of participants: Group1: 100 lung cancer patients scheduled for surgery resection of lung cancer. Group2: 100 high-risk healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of the proteomic and volatolomic signature in samples of respiratory exhalation, serum, and urine from patients with lung cancer (stage I/II) and healthy individuals at high risk. | 12 months
  Enrolling two cohorts at baseline: healthy individuals at high risk with negative LDCT (no suspicious oncological findings) vs. patients with early-stage I/II lung cancer candidates for surgical resection; sampling in lung cancer patients will be performed pre-intervention. We will assess and compare the serum and urinary proteomic and volatile organic compound profiles, serum and respiratory, of the two cohorts under study at baseline and changes in proteomic and volatile organic compound signature at 12 months from baseline.

SECONDARY OUTCOMES:
Omics-Data intagration. | 6 months
  The serum proteomic and serum volatomomic, urinary, and respiratory data will be compared using algorithms based on artificial intelligence and deep learning. Data from each test, including patient follow-up, will be analyzed using multivariate statistical analysis of samples with multivariable logistic and Cox proportional hazards regression models to identify the most significant variables.

CONTACTS AND LOCATIONS:
Locations (1):
- Europen insitute of Oncology- Division of Thoracic Surgery, Milan, Italy